CLINICAL TRIAL: NCT06160024
Title: Data Quality of National Quality Indicators in Long-term Care Facilities: a Validation and Evaluation Study (NIP-Q-UPGRADE Sub-aim 1.4 and 1.9)
Brief Title: Data Quality of National Quality Indicators in Long-term Care Facilities: a Validation and Evaluation Study
Acronym: NIP-Q-UPGRADE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University of Applied Sciences and Arts of Southern Switzerland (Other); Institut et Haute Ecole de la Santé la Source (Other)
Responsible Party: Principal Investigator, Franziska Zúñiga, Principal Investigator, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: WP 1.4_1.9
Record Dates: First submitted 2023-11-12; First posted 2023-12-07 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Reliability of National Quality Indicator Data

STUDY DESIGN:
Intervention Model Description: The study addresses long-term care facilities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long-term care facilities (Other): All participating facilities will be offered the same bundle of measures, with core and optional or adaptable components based on the identified needs.
  Interventions: Behavioral: Program to improve data quality of national quality indicators

INTERVENTIONS:
Behavioral: Program to improve data quality of national quality indicators — Interventions will be developed based on the findings from the first data collection period.
  A bundle of interventions (Program to improve data quality of national quality indicators) will be offered to participating long-term care facilities to support changing behavior in data collection procedures via training and supporting material as implementation strategies with the goal to improve the data quality of the national quality indicators. The program will be tested in a separate pilot study. The second data collection period in the current study will be used to evaluate the effect of the implemented program.

SUMMARY:
This multiple-methods study with two data collection points (T0 and T1) aims to:

1. assess inter-rater reliability of the six national quality indicators in long-term care facilities (LTCFs) for older people in Switzerland (T0);
2. explore determinants of data quality of the national quality indicators (T0),
3. evaluate adoption and effectiveness of a bundle of measures to improve data quality of the national quality indicators (T1).

The study will take place in three language regions of Switzerland. The intended sample is 30 LTCFs . The current reliability of the national quality indicator data will be assessed by comparing two independent quality indicator assessments for the same 30 residents per facility. Afterwards a focus group discussion will be conducted in each facility to explore determinants (barriers and facilitators) to data collection of the national quality indicators. Findings from the first data collection period will be used to develop a program with a bundle of measures (interventions and implementation strategies) to improve data quality of the national quality indicators. The program will be piloted in a separate study and then implemented in the LTCFs, which took part in the initial data collection. The second data collection period will start 3 months after the implementation of the program. A survey of healthcare and management staff will be conducted to assess implementation outcomes. A second reliability assessment of the quality indicators will be conducted with the same procedures to evaluate the effectiveness of the implemented measures.

DETAILED DESCRIPTION:
This multicentre study uses a multi-method approach to assess current data quality of the national quality indicators in Swiss LTCFs and to evaluate a program with a bundle of measures designed to improve data quality of these quality indicators. The study aims to recruit a convenience sample of 30 LTCFs in three language regions (18 German speaking, 9 French speaking and 3 Italian speaking).

The study will use 2 data collection time points, T0 in 2023 and T1 in 2025. Between the two data collections a program with bundle of measures to improve the data quality of the national quality indicators data will be developed and implemented in the participating facilities. The study will use the following procedures:

1. Assessment of the reliability of the national quality indicators data in LTCFs:

   For each participating facility, a double collection of the quality indicators data will be carried out for 30 consecutive assessments of residents over a period of up to 6 months (duration depends on the size of the LTCF, each resident has a needs assessment at least every 180 days, during which quality indicator data are assessed routinely). One professional from each LTCF will be specifically trained in data collection by the research team and will carry out gold standard assessments. Other nursing staff members will conduct the assessments as part of the usual care process. The trained assessor will conduct the assessments of the quality indicators for the same residents in the same assessment period independently, whenever possible based on the electronic health record of the resident, in case of self-reported pain residents may be asked directly, if the data is not recorded daily with a protocol. The data will be entered in a secure online electronic data collection platform (REDCap). An administrative staff member will extract data from routine assessments to enter it in REDCap and the trained assessor will register the gold standard assessment him-/herself. Monthly online monitoring meetings will be conducted with the trained assessors to discuss any difficulties in the assessments and ensure adherence to study procedures.
2. Exploration of the determinants of data quality:

   A focus group discussion with 4-6 staff members involved in organising and conducting the data collection or quality assurance of the quality indicators data i.e., registered nurses or licensed practical nurses, quality managers, will be conducted in each facility after the data collection to assess data reliability is finished. Observed problems concerning data reliability will be discussed to elicit possible sources of errors as well as factors facilitating or hindering correct data collection. The focus group will last around 1h.
3. Evaluation of adoption and effectiveness of a bundle of measures to improve the national quality indicator data will be collected starting three months after implementation of the developed measures.

An online survey of LTCF staff members will be conducted to assess adoption of the intervention components. Eligible to participate will be all facility staff members who were involved in or affected by the introduced data quality improvement measures. To assess effectiveness, inter-rater reliability assessment will be performed in the same way as in aim 1. Effectiveness is defined as an improvement in inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

Long-term care facilities:

* have cantonal recognition as an inpatient long-term care facility
* work with nationally recognized standardized assessment instruments (i.e., RAI-NH, BESA or Plaisir/Plex)
* have at least 30 long-term residents
* have at least two different internal staff members who are involved in the data collection for the national quality indicators
* are willing to participate in two data collections (2023 and 2025) and in between to implement a implement a package of measures to optimise the reliability of the data for the national quality indicators.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of agreement on the presence of malnutrition | up to 6 months at each time point
  Agreement on weight loss of 5% or more in the last 30 days or of 10% or more in the last 180 days per resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the presence of self-reported pain | up to 6 months at each time point
  Agreement on presence of daily moderate or higher pain intensity or with non-daily very strong pain intensity in the last 7 days per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the presence of observed pain | up to 6 months at each time point
  Agreement on presence of daily moderate or higher pain intensity or non-daily very strong pain intensity in the last 7 days per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the presence of trunk fixation or seating that prevents the resident from rising | up to 6 months at each time point
  Agreement on presence of daily fixation of the trunk or with seating that prevented the resident from rising in the last 7 days per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the presence of bedrails | up to 6 months at each time point
  Agreement on presence of daily use of bedrails or other devices on all open sides of the bed that did not allow the resident to leave the bed independently in the last 7 days per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators
Change in the rate of agreement on the presence of polypharmacy | up to 6 months at each time point
  Agreement on presence of 9 or more active ingredients in the last 7 days per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the level of cognitive impairment | up to 6 months at each time point
  Agreement on score on the Cognitive Performance Scale per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the presence of depression | up to 6 months at each time point
  Agreement on score on the Depression Rating Scale per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Change in the rate of agreement on the assessment of life expectancy | up to 6 months at each time point
  Agreement on life expectancy (six months or longer, less than six months or not clarified) per assessed resident between routine assessor and gold standard assessor.
  Primary effectiveness outcomes include all 6 quality indicators and 3 variables used for risk adjustment of quality indicators.
Primary implementation outcome: The rates of adoption of the intervention components of the program to improve the data quality of the national quality indicators | within 8 weeks
  The program with the intervention components will be defined after the first data collection period and will include training and supporting materials

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Zúñiga, Prof. Dr., Principal Investigator — University of Basel
Locations (3):
- Switzerland (3):
  - Institut für Pflegewissenschaft - Nursing Science (INS), University of Basel, Basel, Basel
  - Institut et Haute Ecole de la Santé La Source, Lausanne, Canton of Vaud
  - Scuola universitaria professionale della Svizzera italiana, Manno, Canton Ticino